CLINICAL TRIAL: NCT03758664
Title: A Phase I/IIa, Multicenter, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics of ICP-192 in Patients With Advanced Solid Malignancies
Brief Title: Clinical Study of ICP-192 in Solid Tumors Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00301
Record Dates: First submitted 2018-11-22; First posted 2018-11-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor
Keywords: FGFR gene abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-192 (Experimental): The initial dose of ICP-192 is 2 mg, QD, and dose escalation schedule may be modified based on the safety and PK from the previous dose. Tentatively seven dose levels will be evaluated.
  Interventions: Drug: ICP-192

INTERVENTIONS:
Drug: ICP-192 — Drug: ICP-192 Dose levels will be escalated following accelerated titration and modified "3+3" dose escalation scheme,

SUMMARY:
Open-label, non-randomized, Phase I/IIa, dose-escalating, dose-extension, first-in-man study.

DETAILED DESCRIPTION:
The study consisted of a screening period, a treatment period with 21 days of repeated treatment per cycle (duration treatment with ICP-192), and a follow-up period (28 days after last dose). The recruited patients receive a single dose on day 1, then after a 3-day washout period, repeated dosing will be followed. The starting dose is 2 mg, QD, and dose escalation will follow accelerated titration and modified 3+3 dose-finding schema. The dose-limiting toxicity (DLT) assessment period consisted of Cycle 0 (single dose and washout period) and Cycle 1 (21-day cycle).

ELIGIBILITY:
Inclusion Criteria:

1. An unresectable or metastatic advanced malignant solid tumor confirmed by histopathology that has failed to respond to known treatment or has recurred;Subjects who progress under standard treatment, are intolerant to standard treatment, or do not have standard treatment (dose escalation phase)
2. Tissue or cell pathology confirmed unresectable, recurrent or metastatic (AJCC version 8 TNM staging IV (2017), biliary tract malignant tumor, or intolerance to first-line chemotherapy failure (twice (defined as reduction still cannot tolerate) first-line chemotherapy, neoadjuvant/progress/adjuvant chemotherapy after 6 months recurrence can be selected (dose extension stage); - At least one evaluable disease according to RECIST1.1
3. FGFR2 translocation/fusion has been reported or FGFR2 translocation/fusion has been detected in central laboratory (dose extension phase);
4. Age ≥18 and ≤75
5. There is at least one evaluable lesion according to RECIST1.1 criteria
6. ECOG strength score is 0-1 (dose escalation stage), and ECOG strength score is 0-2 (dose expansion stage).
7. The expected survival time is more than 3 months
8. The organ function level must meet the following requirements (subject to the upper limit of normal value in the clinical trial center):

   A) bone marrow: absolute count of neutrophils (ANC)≥1.5*109/L (1500/mm3), platelet ≥75*109/L, hemoglobin ≥9g/dL; B) coagulation function: international standardized ratio of prothrombin time and partial thrombin time <1.5 times the upper limit of normal value; C) liver: serum bilirubin ≤1.5 times the upper limit of normal value (tumor involvement in the liver ≤2.5 times the upper limit of normal value), aspartic aminotransferase (AST) and alanine aminotransferase (ALT)≤3 times the upper limit of normal value (AST and ALT≤5 times the upper limit of normal value in the case of liver metastasis); D) serum creatinine ≤1.5 times the upper limit of normal value, or creatinine clearance ≥70mL/min (calculated according to the Cockroft-gult formula).
9. Volunteer to enroll and sign informed consent to follow the treatment protocol and visit plan.

Exclusion Criteria:

* Previous treatment with FGFR small molecule inhibitors or antibody drugs.
* Anti-cancer therapy, such as chemotherapy (except for oral fluorouracil), immunotherapy, hormonal, targeted therapy, or investigational agents within four weeks of the first dose of ICP-192, oral fluorouracil agents within two weeks of the first dose of ICP-192.
* Major surgery within 6 weeks of the first dose of ICP-192.
* Blood phosphate persistently above ULN with intervene therapy within two weeks of the first dose of ICP-192.
* Significant GI disorder(s) that could interfere with the absorption, metabolism, or excretion of ICP-192.
* Central nervous system (CNS) metastasis
* Current clinically significant cardiovascular disease including:
* Any class 3 or 4 cardiac disease such as arrhythmia, congestive heart failure or myocardial infarction defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) < 50%, Primary cardiomyopathy, clinical significant QTc prolong history or QTc>470ms (female) QTc>450ms (male)
* Known active bleeding within 2 months of screening or 6 months of bleeding history.
* According to the investigator's judgement, there are evidences of a serious or uncontrollable systemic disease (such as unstable or uncompensated respiratory, liver or kidney disease); or any unstable systemic disease (including active clinically serious infections, uncontrolled hypertension, liver and kidney or metabolic diseases)
* History of interstitial pneumonia, deep vein thrombosis, pulmonary embolism. Stroke or intracranial hemorrhage within 6 months before the first dose of ICP-192.
* History of organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Any corneal or retinal abnormalities that may increase ocular toxicity, including but not limited to:
* History of central serous retinopathy (CSR) or retinal vein occlusion (RVO) disease or has related diseases;
* Active age-related macular degeneration (AMD);
* Diabetic retinopathy with macular edema;
* Uncontrollable glaucoma;
* Keratonosus, such as Keratitis, keratoconjunctivitis, keratopathy, corneal wear, inflammation or ulceration.
* Known active infection with HBV, HCV or HIV or any uncontrolled active systemic infection
* Any toxicities must recover to ≤ Grade 1 from prior anti-cancer therapy (excluding alopecia, nausea and vomiting).
* Lactating or pregnant women, or women who will not use contraception during the study and for 180 days after the last dose of study drug if sexually active and able to bear children.
* Investigators believe that the patients are not eligible for enrollment for the other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events(Phase 1 dose escalation) | From the time a signed and dated ICF until 28 days after last dose of study drug
  Adverse events graded by CTCAE V5.0 as a measurement of the safety and tolerability profile of ICP-192
Objective Response Rate(ORR)(Phase 2a dose expansion) | At the end of Cycle 4(each cycle is 21 days)
  Objective response based on assessment of confirmed Complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST).

SECONDARY OUTCOMES:
Cmax | At the end of Cycle 1(each cycle is 21 days)
  Single dose PK parameters include the peak plasma concentration (Cmax)
AUC | At the end of Cycle 1(each cycle is 21 days)
  Area under the plasma concentration vs. time curve (AUC)
Apparent half-life for designated elimination phases (t½) | At the end of Cycle 1(each cycle is 21 days)
  will be measured and calculated with noncompartmental analysis using WinNonlin
Food effect | Day 1 - 6 after single dose
  ICP-192 concentrations in plasma and urine after dosing in fed and fasted condition
Objective Response Rate(ORR) (Phase 1 dose escalation) | At the end of Cycle 4(each cycle is 21 days)
  Objective response based on assessment of confirmed Complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST).
Disease control rate(DCR) | At the end of Cycle 4(each cycle is 21 days)
  DCR based on assessment of confirmed Complete response (CR), partial response (PR) or stable disease(SD) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST).
Duration of Objective Response (DOR) | At the end of Cycle 4(each cycle is 21 days)
  Duration of objective response is time interval from the first date that criteria for complete response or partial response are met to the first date of progression of disease
Progression Free Survival (PFS) | At the end of Cycle 4(each cycle is 21 days)
  Progression free survival is the time period from start of study medication till the disease progression or death, whichever occurs first.
Correlationship between FGFR aberrations with efficacy. (Phase 2a dose expansion) | At the end of Cycle 4(each cycle is 21 days)
  Correlationship between FGFR mutation/refusion with ORR

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Shanghai East Hospital
Locations (7):
- China (7):
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan cancer hospital & Affiliated Tumor Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan cancer hospital & the affiliated cancer hospital of xiangya school of medicine ,central south university, Changsha, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Cancer hospital of the university of Chinese academy of sciences, Hangzhou, Zhejiang